CLINICAL TRIAL: NCT06982690
Title: Impact of Anesthesia Modality on Recurrence and Progression in High-Risk Non-Muscle Invasive Bladder Cancer: A Randomized Controlled Trial Comparing Spinal Versus General Anesthesia
Brief Title: Anesthesia Modality and Oncologic Outcomes in High-Risk NMIBC: A Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Director, Department of Urology at National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202411115RINE
Record Dates: First submitted 2025-04-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: NMIBC; TURBT; Bladder (Urothelial, Transitional Cell) Cancer; Bladder Cancer Recurrence; Anesthesia, General; Anesthesia,Spinal
Keywords: bladder cancer; general anesthesia; spinal anesthesia; recurrence; TURBT
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Neoplasms; Urinary Bladder Neoplasms; Recurrence | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Anesthesia (Placebo Comparator)
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia (Active Comparator)
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — A total of 10-12 mg of 0.5% bupivacaine will be administered into the cerebrospinal fluid of the subarachnoid space using a 25-gauge Quincke spinal needle via an 18-gauge introducer (adjusted by body height). Midazolam (2-5 mg) may be used to decrease anxiety.
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — Induction will be performed with propofol (0.5-1.5 mg/kg) and fentanyl (1-2 µg/kg), and anesthesia will be maintained with sevoflurane (1-3 vol %) via a laryngeal mask or endotracheal intubation. Rocuronium (0.5-0.6 mg/kg) will be used for induction, maintenance and occurrence of obturator jerk.
  Arms: General Anesthesia

SUMMARY:
To demonstrate the superior efficacy of spinal anesthesia (SA) versus general anesthesia (GA) according to the delay of time to recurrence in high-risk NMIBC patients up to Week 104 after TURBT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years for male subjects or postmenopausal female subjects
* ECOG performance status 0-2
* Patients with suspected or newly diagnosed UBUC
* ASA I or II
* Patients with any other adequately treated Stage I or II cancer except UC, from which the subject has been disease free for 5 years
* Adequate renal function, defined as a serum creatinine (Cre) concentration ≤ the institutional ULN
* Adequate hepatic function, defined as total bilirubin ≤ the institutional ULN and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ the institutional upper limit of normal (ULN)

Exclusion Criteria:

* Patients with prior or concurrent UC involving the renal pelvis, ureter or urethra
* Patients with clinical evidence of MIBC or mUC
* Immunocompromised or immunosuppressed patients
* Patients with chronic use of anti-inflammatory agents or beta-blockers
* Patients with difficult airways or other significant cardiovascular comorbidities (severe aortic stenosis, significant pulmonary disease, CHF) who are intolerant to GA
* Patients with elevated intracranial pressure (ICP), primarily due to intracranial mass and trauma or infection at the site of SA
* Patients with a serious uncontrolled medical disorder (e.g., trauma, fracture) or active infection that would impair their ability to receive spinal or GA
* Patients with known allergies to propofol, fentanyl, sevoflurane, or bupivacaine
* Subjects with a known history or family history of malignant hyperthermia
* Subjects with bleeding diathesis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence in high risk NMIBC patients | From date of TURBT (Study Day 0) until documented recurrence or last follow-up, up to 104 weeks
  The time to recurrence is defined as the number of days from TURBT to the day on which the subject presents with gross hematuria, positive urine cytology, all-risk bladder tumor relapse or newly diagnosed upper tract UC with pathological confirmation, radiographically detected tumor metastasis, or cancer-specific death beyond 90 days after diagnosis, whichever occurs first.

SECONDARY OUTCOMES:
Time to event in high-risk NMIBC patients up to Week 104 | From date of TURBT (Study Day 0) until documented recurrence or last follow-up, up to 104 weeks
  An event is defined as a composite variable reflecting the recurrence of a high-risk disease (any high-grade disease, any T1 tumor, multifocal disease, >3 cm, variant histology, lymphovascular invasion, or CIS), disease progression or metastasis, BCG unresponsiveness, or cancer-specific death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, College of Medicine, National Taiwan University, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fang CW, Shau WY, Fan SZ, Chueh JS. Comparison of spinal versus general anaesthesia in high-risk non-muscle invasive bladder cancer: study protocol for a randomised controlled trial. BMJ Open. 2025 Nov 28;15(11):e107824. doi: 10.1136/bmjopen-2025-107824. PMID 41314851